CLINICAL TRIAL: NCT01605435
Title: Ghrelin In Frail Elderly Subcutaneous Dose Finding Study
Brief Title: Ghrelin Dose Finding In Frail Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Anne Cappola, Associate Professor of Medicine, University of Pennsylvania
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB 814309
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Results first posted 2018-10-10 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-11

CONDITIONS: The Frailty Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ghrelin Group 1 (Experimental): Dose finding with each of the first two participant coming to the CTRC for four visits greater than or equal to 72 hours apart and on each receiving subcutaneous injection of - placebo (first visit) and three escalating doses of ghrelin 2ug/kg (second visit) , 5 ug/kg (third visit), and 10 ug/kg (fourth visit).
  Interventions: Drug: Ghrelin Group 1
- Ghrelin Group 2 (Experimental): Dose finding with each of the final three participant coming to the CTRC for four visits greater than or equal to 72 hours apart and on each receiving subcutaneous injection of - placebo (first visit) and three escalating doses of ghrelin 5ug/kg (second visit) , 7.5 ug/kg (third visit), and 10 ug/kg (fourth visit).
  Interventions: Drug: Ghrelin Group 2

INTERVENTIONS:
Drug: Ghrelin Group 1 — The first two participants received placebo at baseline visit, 2 mcg/kg as a single subcutaneous dose at Visit 2, 5 mcg/kg as a single subcutaneous dose at Visit 3, and 10 mcg/Kg as a single subcutaneous dose at visit 4. There was 3-10 days between visits.
  Other Names: First dose escalation group
  Arms: Ghrelin Group 1
Drug: Ghrelin Group 2 — The next three participants received placebo at baseline visit, 5 mcg/kg as a single subcutaneous dose at Visit 2, 7.5 mcg/kg as a single subcutaneous dose at Visit 3, and 10 mcg/Kg as a single subcutaneous dose at visit 4.
  Other Names: Second dose escalation group
  Arms: Ghrelin Group 2

SUMMARY:
Frailty is a geriatric syndrome leading to physical deterioration including muscle wasting (sarcopenia) and unintentional weight loss. There are currently no approved therapies for frailty. Ghrelin is a hormone produced by the stomach that stimulates appetite centers in the brain. The purpose of this study is to determine the optimal subcutaneous ghrelin dose as a potential intervention for frail elderly individuals. We will examine food intake and metabolic parameters after placebo and ghrelin administration at three escalating subcutaneously administered doses.

DETAILED DESCRIPTION:
This study is to determine the optimal ghrelin dose for use in a daily subcutaneous dosing study in frail individuals. Using data from our previous study and the published literature, we have designed a single blind, single dose administration study in which we will examine food intake after ghrelin administration and metabolic parameters (plasma glucose, insulin, free fatty acids, and cortisol) pre and post ghrelin administration.We have selected a dose range using our own and previously published studies from which we will determine subcutaneous doses to use in subsequent studies. The selection criteria for subsequent studies will be the dose that maximizes food intake by more than 30% without inducing hyperglycemia or raising cortisol levels. Participants must meet all inclusion criteria and have no exclusion criteria. Data will be analyzed after the first three participants have completed the protocol and used to inform dose modifications for the next three participants. Data from this portion of the study will be analyzed immediately after its completion, to allow updates to the design of the next study.

ELIGIBILITY:
Inclusion Criteria:

* We will include men and women aged 70 or older who are able to provide informed consent and are frail by the Fried criteria (Table 1).
* Table 1. Frailty criteria. Individuals with three, four, or all five criteria are frail.
* Weight loss: Unintentional weight loss of >5% over the previous year

Exhaustion: Two statements are read:

* I felt that everything I did was an effort
* I could not get going. The question is asked "How often in the last week did you feel this way?" 0 = rarely or none of the time (<1 day), 1 = some or a little of the time (1-2 days), 2 = a moderate amount of the time (3-4 days), or 3 = most of the time. A "2" or "3" response to either question is a positive response.

  * Low physical activity: Kcal/week of physical activity calculated from the short version of the Minnesota Leisure Time Activity questionnaire.40 < 383 kcals in men or < 270 kcals/wk in women is positive for this criterion.
  * Slow walking speed: A usual pace, 15-ft walk timed from a defined standing start. For men ≤173 cm tall and women ≤159 cm, ≥7 sec, and for men >173 cm and women > 159 cm, ≥ 6 sec is positive for this criterion.
  * Weakness: Hand grip strength measured with a dynamometer. The average of three measurements performed in the dominant hand is used. For men with BMI ≤ 24 kg/m2, the cutoff is ≤ 29 kg, for BMI 24.1 to 26 the cutoff is ≤ 30 kg, for BMI 26.1 to 28 the cutoff is ≤30 kg, and for BMI > 28 the cutoff is ≤ 32 kg. For women with BMI ≤ 23 kg/m2, the cutoff is ≤ 17 kg, for BMI 23.1 to 26 the cutoff is ≤ 17.3 kg, for BMI 26.1 to 29 the cutoff is ≤ 18 kg, and for BMI > 29 the cutoff is ≤ 21 kg for a positive criterion.

Exclusion Criteria:

1. Diabetes mellitus or fasting glucose ≥ 126 mg/dL
2. Hospitalization for stroke, myocardial infarction, coronary artery bypass graft surgery, vascular surgery in the past six months.
3. NYHA Class III or IV congestive heart failure
4. Therapy for cancer in the past 12 months, except non-melanoma skin cancer
5. BMI≥ 30 kg/m2
6. Current use of corticosteroids other than topical, ophthalmic, and inhaled preparations
7. Therapy with megestrol acetate or dronabinol within the last 6 weeks
8. TSH measured as <0.4 mU/L or greater than 10mU/L
9. Abnormal liver function tests (LFTs > 2x upper limit of normal)
10. Hemoglobin < 11g/dL
11. Insulin-like growth factor-I (IGF-I) above the age-specific reference range
12. History of surgery within the last 30 days
13. Unstable medical or psychological conditions or unstable home or food environment
14. Cognitive deficit as defined by a Folstein Mini Mental State Exam score < 18/30
15. Depression (defined as a score of >11 on the Geriatric Depression Questionnaire)

    -

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne R. Cappola, M.D., Sc.M., Principal Investigator — University Of Pennsylvania, Perelman School of Medicine, Department of Endocrinology, Diabetes and Metabolism
Locations (1):
- Clinical and Translational Research Center, University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from community dwelling adults meeting study criteria expressing interest in participating in research studies at University of Pennsylvania.
Pre-assignment Details: Dose finding with each participant receiving placebo at their first study visits and three escalating doses of ghrelin, separated by 3-7 days in visits 2,3 and 4.
Groups:
- Initial Dosing Group: Visit 1: Placebo Visit 2: 2 ug/kg ghrelin Visit 3: 5 ug/kg ghrelin Visit 4: 10 ug/kg ghrelin
- Second Dosing Group: Visit 1: Placebo Visit 2: 5 ug/kg ghrelin Visit 3: 7.5 ug/kg ghrelin Visit 4: 10 ug/kg ghrelin
Period: Overall Study
Arm/Group | Initial Dosing Group | Second Dosing Group
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ghrelin: Dose finding with each participant receiving placebo and three doses of ghrelin, separated by 3-7 days
  Ghrelin: The first three participants will receive 2 mcg/kg as a single subcutaneous dose at Visit 3, 5 mcg/kg as a single subcutaneous dose at Visit 4, and 10 mcg/Kg as a single subcutaneous dose at visit 5. There will be 3-10 days between visits. The next three participants will receive either the same dosing at the first three, a regimen that includes an intermediate dose (e.g., 7.5 mcg/kg), or higher (e.g., 12, 15, and 18 mcg/kg) doses.
Arm/Group | Ghrelin
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years] | 85 [79 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Treatment Emergent Adverse Events
Description: Number and type of treatment emergent adverse events
Time Frame: 30 days following the last administration of study treatment.
Population: At the first visit all participants received s.c. placebo. The first two participants received 2 ,5, and 10ug/kg of ghrelin at visit 2,3 and 4 consecutively. The final three participants received 5,7.5, and 10ug/kg of s.c. ghrelin at visits 2,3 and 4 consecutively.
Measure: Number; unit: Events
Groups:
- Placebo: All 5 subjects received s.c. placebo at visit 1.
- 2ug/kg: The first two participants received 2ug/kg of s.c. ghrelin at visit 2.
- 5ug/kg: The first two participants received 5ug/kg of s.c. ghrelin at visit 3. The final three participants received 5ug/kg of s.c. ghrelin at visits 2.
- 7.5ug/kg: The final three participants received 7.5ug/kg of s.c. ghrelin at visit 3.
- 10ug/kg: The first two participants received 10ug/kg of s.c. ghrelin at visit 4. The final three participants received 10ug/kg of s.c. ghrelin at visit 4.
Arm/Group | Placebo | 2ug/kg | 5ug/kg | 7.5ug/kg | 10ug/kg
Number analyzed (Participants) | 5 | 2 | 5 | 3 | 5
Events
  burping | 1 | 0 | 1 | 0 | 0
  sensation of warmth | 0 | 0 | 0 | 2 | 1
  bristley feeling | 1 | 0 | 0 | 0 | 0
  dizzy | 0 | 0 | 0 | 1 | 0
  awareness of old incision | 0 | 0 | 0 | 1 | 0
  euphoria | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Median Energy Intake
Description: Median energy intake at breakfast, which was served 30 minutes post-placebo or ghrelin administration demonstrated at each dose level.
Time Frame: 30 mins post-ghrelin or placebo
Population: At the first visit all participants received s.c. placebo. The first two participants received 2 ,5, and 10ug/kg of ghrelin at visit 2, 3 and 4 consecutively. The final three participants received 5,7.5, and 10ug/kg of s.c. ghrelin at visits 2,3 and 4 consecutively.
Measure: Median (Full Range); unit: Kilocalories
Groups:
- 2 mcg/kg: The first two participants received 2ug/kg of s.c. ghrelin at visit 2.
- 5mcg/kg: The first two participants received 5ug/kg of s.c. ghrelin at visit 3. The final three participants received 5ug/kg of s.c. ghrelin at visits 2.
- 7.5mcg/kg: The final three participants received 7.5ug/kg of s.c. ghrelin at visit 3.
- 10mcg/kg: The first two participants received 10ug/kg of s.c. ghrelin at visit 4. The final three participants received 10ug/kg of s.c. ghrelin at visit 4.
Arm/Group | Placebo | 2 mcg/kg | 5mcg/kg | 7.5mcg/kg | 10mcg/kg
Number analyzed (Participants) | 5 | 2 | 5 | 3 | 5
Kilocalories | 535.16 [482.14 to 670.05] | 578 [436.28 to 719.872] | 813 [500.87 to 1083.75] | 852 [790.26 to 917.69] | 862.04 [493.34 to 925.91]

3. Primary Outcome: Percentage of Total Energy Intake Relative to Placebo
Description: % of total energy relative to placebo - breakfast served 30 minutes post-placebo or ghrelin administration.
Time Frame: 30 mins post-ghrelin or placebo
Population: as for outcome 1
Measure: Number; unit: percentage of placebo intake
Arm/Group | Placebo | 2 mcg/kg | 5mcg/kg | 7.5mcg/kg | 10mcg/kg
Number analyzed (Participants) | 5 | 2 | 5 | 3 | 5
percentage of placebo intake | 100 | 110 | 135 | 139 | 129

4. Primary Outcome: Growth Hormone
Description: median growth hormone peak 30 minutes after placebo/ghrelin.
Time Frame: 30 minutes after ghrelin administration
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Groups:
- 2mcg/kg: The first two participants received 2ug/kg of s.c. ghrelin at visit 2.
Arm/Group | Placebo | 2mcg/kg | 5mcg/kg | 7.5mcg/kg | 10mcg/kg
Number analyzed (Participants) | 5 | 2 | 5 | 3 | 5
ng/mL | 3.71 [2.52 to 5.91] | 16.87 [4.27 to 29.47] | 31.81 [7.85 to 50.00] | 39.20 [12.20 to 39.21] | 33.63 [4.99 to 50.00]

5. Primary Outcome: Cortisol Level
Description: Cortisol response to ghrelin or placebo - levels at 0, 60 and 120 minutes after dosing
Time Frame: 0, 60 and 120 minutes after dosing
Population: as for outcome 1
Measure: Median (Full Range); unit: mcg/dL
Arm/Group | Placebo | 2ug/kg | 5ug/kg | 7.5ug/kg | 10ug/kg
Number analyzed (Participants) | 5 | 2 | 5 | 3 | 5
mcg/dL
  0 minutes, baseline | 26.4 [19.3 to 35.2] | 27.1 [24.5 to 29.7] | 28.4 [20.6 to 30.4] | 21.5 [20.7 to 28.6] | 22.7 [20 to 30.9]
  60 minutes after dosing | 18.6 [14.7 to 22.6] | 22.0 [21.2 to 22.8] | 35.3 [18.4 to 42.7] | 33.7 [16.2 to 36.0] | 31.8 [18.2 to 41.1]
  120 minutes after dosing | 18.8 [16.8 to 32.8] | 29.7 [29 to 30.4] | 27.5 [19.0 to 37.7] | 32.5 [17.9 to 33.0] | 26.4 [20.5 to 30.9]

6. Primary Outcome: Glucose Levels
Description: Median fasting and peak postprandial Glucose levels (60 or 90 minutes from dosing) at placebo and at each ghrelin dose.
Time Frame: 0 minutes (baseline) and 60 or 90 minutes from dosing
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Placebo | 2mcg/kg | 5mcg/kg | 7.5mcg/kg | 10mcg/kg
Number analyzed (Participants) | 5 | 2 | 5 | 3 | 5
mg/dL
  Fasting (0 minutes) | 93 [89 to 122] | 90 [87 to 93] | 91 [88 to 102] | 104 [89 to 113] | 94 [88 to 106]
  peak postprandial (60 or 90 minutes after dosing) | 142 [125 to 166] | 141 [135 to 146] | 162 [145 to 187] | 167 [147 to 196] | 164 [153 to 184]

7. Primary Outcome: Insulin Level
Description: Median fasting insulin levels at baseline and 90 minutes after dosing
Time Frame: 0 and 90 minutes after dosing
Population: as for outcome 1
Measure: Median (Full Range); unit: uIU/mL
Arm/Group | Placebo | 2ug/kg | 5ug/kg | 7.5ug/kg | 10ug/kg
Number analyzed (Participants) | 5 | 2 | 5 | 3 | 5
uIU/mL
  Fasting (0 minutes) | 12.9 [2.0 to 16.0] | 14.8 [13.0 to 16.5] | 8.5 [3.1 to 16.0] | 8.7 [7.0 to 17.2] | 9.7 [4.7 to 16.9]
  90 minutes after dosing | 82.9 [12.9 to 164.5] | 115.8 [76.5 to 155.0] | 109.5 [60.1 to 186.5] | 77.6 [38.9 to 149.0] | 85.8 [38.8 to 186.5]

8. Primary Outcome: Free Fatty Acid Level
Description: Free Fatty Acid levels (mEq/L) at 60 and 90 minutes after meal (90 and 120 minutes)
Time Frame: 90 and 120 minutes after dosing
Population: as for outcome 1
Measure: Median (Full Range); unit: mEq/L
Arm/Group | Placebo | 2mcg/kg | 5mcg/kg | 7.5mcg/kg | 10mcg/kg
Number analyzed (Participants) | 5 | 2 | 5 | 3 | 5
mEq/L
  90 minutes | 0.17 [0.12 to 0.35] | 0.11 [0.10 to 0.12] | 0.22 [0.09 to 0.42] | 0.35 [0.20 to 0.46] | 0.29 [0.08 to 0.36]
  120 minutes | 0.10 [0.06 to 0.12] | 0.08 [0.05 to 0.11] | 0.09 [0.04 to 0.27] | 0.14 [0.11 to 0.15] | 0.12 [0.06 to 0.14]

ADVERSE EVENTS:
Time Frame: Recorded from study screen through 30 days after the final study visit. Assessed systematically during study visits at time 0, 15, 30, 45, 60, 90 120, and 150 minutes after dosing and 1 day after all study visits by telephone call to subject.
Groups:
- Placebo: Visit 1 for all five subjects placebo injected s.c. at time 0
- 2mcg/kg: Visit 2 for the first two subjects 2mcg/kg ghrelin injected s.c at time 0
- 5mcg/kg: Visit 3 for the first two subjects Visit 2 for the last three subjects 5mcg/kg ghrelin injected s.c. at time 0
- 7.5mcg/kg: Visit 3 for the last three subjects 7.5mcg/kg ghrelin injected at time 0
- 10mcg/kg: Visit 4 for all five subjects
Arm/Group | Placebo | 2mcg/kg | 5mcg/kg | 7.5mcg/kg | 10mcg/kg
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2 | 0/5 | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 2/5 | 0/2 | 1/5 | 3/3 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=5) | 2mcg/kg (N=2) | 5mcg/kg (N=5) | 7.5mcg/kg (N=3) | 10mcg/kg (N=5)
bristley feeling in chest (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — reported day after placebo visit, occurred and resolved in one minute with no action.
awareness of sternotomy incision (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — occurred during visit 30 minutes after ghrelin administration and resolved within 15 minutes with no action.
dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — "dizzy is too strong - woozy"
burping (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — during study visit 15 minutes after meal completion
warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) — passing sensation between 45 and 60 minutes from ghrelin injection resolving with no action
euphoria (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — passing feeling during study visit 1 hour after ghrelin administration

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No